CLINICAL TRIAL: NCT02557672
Title: Prothrombin Complex Concentrate (PCC) Compared to Fresh Frozen Plasma (FFP) for Post-cardiopulmonary Bypass Coagulopathy and Bleeding, a Prospective Randomized Trial at Large US Medical Center.
Brief Title: PCC vs. FFP for Post Cardiopulmonary Bypass Coagulopathy and Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Gregory A. Nuttall, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-009579
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Bleeding; Blood Loss, Surgical; Cardiovascular Surgical Procedures; Prothrombin Complex Concentrates; Fresh Frozen Plasma
MeSH Terms: conditions — Hemorrhage; Blood Loss, Surgical | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fresh frozen plasma (Active Comparator): After cardiopulmonary bypass, patients will receive protamine at dose 0.01 mg/unit of heparin given with target activated clotting time (ACT) within 10% of baseline value. After protamine administration the ACT, complete blood count (CBC), prothrombin time (PT)/ international normalized ratio (INR), activated partial thromboplastin time (APTT), and fibrinogen, will be collected via preexisting arterial access. If ACT >10% baseline additional protamine will be given at the anesthesiologists discretion. Evaluation and determination of excessive microvascular bleeding in the surgical field will occur 10 minutes after return of ACT to within 10% of baseline. Patients with clinical evidence of excessive microvascular bleeding in the surgical field as determined by the surgical team, along with a PT >16.6 sec/ INR >1.6 sec will receive fresh frozen plasma as this is standard therapy per our institutional algorithm at a dose of 10-15 mL/kg rounded up to the nearest unit.
  Interventions: Biological: Fresh frozen plasma (FFP)
- Prothrombin complex concentrate (Experimental): After cardiopulmonary bypass, patients will receive protamine at dose 0.01 mg/unit of heparin given with target ACT within 10% of baseline value. After protamine administration the ACT, CBC, PT/ INR, APTT, and fibrinogen, will be collected via preexisting arterial access. If ACT >10% baseline additional protamine will be given at the anesthesiologists discretion. Evaluation and determination of excessive microvascular bleeding in the surgical field will occur 10 minutes after return of ACT to within 10% of baseline. Patients with clinical evidence of excessive microvascular bleeding in the surgical field as determined by the surgical team, along with a PT >16.6 sec/ INR >1.6 sec will receive Prothrombin complex concentrate (Human) 15 units/kg.
  Interventions: Drug: Prothrombin complex concentrate (Human)

INTERVENTIONS:
Drug: Prothrombin complex concentrate (Human) — PCC (Kcentra)
  Other Names: Kcentra
  Arms: Prothrombin complex concentrate
Biological: Fresh frozen plasma (FFP) — FFP
  Arms: Fresh frozen plasma

SUMMARY:
This will be the first prospective randomized controlled clinical trial directly comparing Prothrombin Complex Concentrate (PCC) Compared to Fresh Frozen Plasma (FFP) for post cardiopulmonary bypass microvascular bleeding and factor-mediated coagulopathy. Is there a difference in bleeding and transfusion requirements in patients received PCC versus FFP?

ELIGIBILITY:
Inclusion Criteria

All subjects accepted for this study must:

* Be 18 years of age
* Be undergoing elective cardiac surgical procedure utilizing cardiopulmonary bypass
* Have evidence of excessive microvascular bleeding in the surgical field as determined by the surgical team in addition to a PT >16.6 sec or INR >1.6 sec.

Exclusion Criteria

Subjects who have one or more of the following will be excluded from the study:

* Are unable to grant informed consent or comply with study procedure
* History of hypercoagulable condition (e.g. Factor V Leiden, AT-3 deficiency, Prothrombin gene mutation, Anti-phospholipid antibody syndrome, etc) or previous unprovoked thromboembolic complications
* Coagulopathic conditions such as factor deficiencies, factor inhibitors, heparin induced thrombocytopenia, or use of intravenous anticoagulants other than heparin at the time of cardiovascular surgery
* Thromboembolic event within past 3 months
* Received oral therapy with clopidogrel, prasugrel, rivaroxaban or dabigatran within the past 5 days
* Patients taking chronic warfarin therapy who have not discontinued treatment and demonstrated an INR <1.3 prior to surgery
* Fibrinogen level <150 mg/dL on initial post cardiopulmonary bypass labs
* Antithrombin 3 level < 80% control (preoperative)
* Are undergoing emergency open heart-surgery
* Cardiopulmonary bypass time is expected to be < 30 minutes
* Age < 18 years of age
* Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Nuttall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnekian V, Camous J, Fattal S, Rezaiguia-Delclaux S, Nottin R, Stephan F. Use of prothrombin complex concentrate for excessive bleeding after cardiac surgery. Interact Cardiovasc Thorac Surg. 2012 Sep;15(3):382-9. doi: 10.1093/icvts/ivs224. Epub 2012 May 23. PMID 22623627
- [Background] Ballotta A, Saleh HZ, El Baghdady HW, Gomaa M, Belloli F, Kandil H, Balbaa Y, Bettini F, Bossone E, Menicanti L, Frigiola A, Bellucci C, Mehta RH. Comparison of early platelet activation in patients undergoing on-pump versus off-pump coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2007 Jul;134(1):132-8. doi: 10.1016/j.jtcvs.2007.01.055. PMID 17599498
- [Background] Demeyere R, Gillardin S, Arnout J, Strengers PF. Comparison of fresh frozen plasma and prothrombin complex concentrate for the reversal of oral anticoagulants in patients undergoing cardiopulmonary bypass surgery: a randomized study. Vox Sang. 2010 Oct;99(3):251-60. doi: 10.1111/j.1423-0410.2010.01339.x. PMID 20840339
- [Background] Ferreira J, DeLosSantos M. The clinical use of prothrombin complex concentrate. J Emerg Med. 2013 Jun;44(6):1201-10. doi: 10.1016/j.jemermed.2012.12.022. Epub 2013 Apr 18. PMID 23602147
- [Background] Goldberg AD, Kor DJ. State of the art management of transfusion-related acute lung injury (TRALI). Curr Pharm Des. 2012;18(22):3273-84. doi: 10.2174/1381612811209023273. PMID 22621274
- [Background] Gorlinger K, Dirkmann D, Hanke AA, Kamler M, Kottenberg E, Thielmann M, Jakob H, Peters J. First-line therapy with coagulation factor concentrates combined with point-of-care coagulation testing is associated with decreased allogeneic blood transfusion in cardiovascular surgery: a retrospective, single-center cohort study. Anesthesiology. 2011 Dec;115(6):1179-91. doi: 10.1097/ALN.0b013e31823497dd. PMID 21970887
- [Background] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381
- [Background] Hanke AA, Joch C, Gorlinger K. Long-term safety and efficacy of a pasteurized nanofiltrated prothrombin complex concentrate (Beriplex P/N): a pharmacovigilance study. Br J Anaesth. 2013 May;110(5):764-72. doi: 10.1093/bja/aes501. Epub 2013 Jan 18. PMID 23335567
- [Background] Holbrook A, Schulman S, Witt DM, Vandvik PO, Fish J, Kovacs MJ, Svensson PJ, Veenstra DL, Crowther M, Guyatt GH. Evidence-based management of anticoagulant therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e152S-e184S. doi: 10.1378/chest.11-2295. PMID 22315259
- [Background] Kaatz S, Kouides PA, Garcia DA, Spyropolous AC, Crowther M, Douketis JD, Chan AK, James A, Moll S, Ortel TL, Van Cott EM, Ansell J. Guidance on the emergent reversal of oral thrombin and factor Xa inhibitors. Am J Hematol. 2012 May;87 Suppl 1:S141-5. doi: 10.1002/ajh.23202. Epub 2012 Apr 4. PMID 22473649
- [Background] Levy JH, Faraoni D, Spring JL, Douketis JD, Samama CM. Managing new oral anticoagulants in the perioperative and intensive care unit setting. Anesthesiology. 2013 Jun;118(6):1466-74. doi: 10.1097/ALN.0b013e318289bcba. PMID 23416382
- [Background] Nuttall GA, Oliver WC, Santrach PJ, Bryant S, Dearani JA, Schaff HV, Ereth MH. Efficacy of a simple intraoperative transfusion algorithm for nonerythrocyte component utilization after cardiopulmonary bypass. Anesthesiology. 2001 May;94(5):773-81; discussion 5A-6A. doi: 10.1097/00000542-200105000-00014. PMID 11388527
- [Background] Pandey S, Vyas GN. Adverse effects of plasma transfusion. Transfusion. 2012 May;52 Suppl 1(Suppl 1):65S-79S. doi: 10.1111/j.1537-2995.2012.03663.x. PMID 22578374
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Thiele RH, Raphael J. A 2014 Update on Coagulation Management for Cardiopulmonary Bypass. Semin Cardiothorac Vasc Anesth. 2014 Jun;18(2):177-89. doi: 10.1177/1089253214534782. PMID 24876232
- [Background] Toy P, Popovsky MA, Abraham E, Ambruso DR, Holness LG, Kopko PM, McFarland JG, Nathens AB, Silliman CC, Stroncek D; National Heart, Lung and Blood Institute Working Group on TRALI. Transfusion-related acute lung injury: definition and review. Crit Care Med. 2005 Apr;33(4):721-6. doi: 10.1097/01.ccm.0000159849.94750.51. PMID 15818095
- [Background] Ortmann E, Besser MW, Sharples LD, Gerrard C, Berman M, Jenkins DP, Klein AA. An exploratory cohort study comparing prothrombin complex concentrate and fresh frozen plasma for the treatment of coagulopathy after complex cardiac surgery. Anesth Analg. 2015 Jul;121(1):26-33. doi: 10.1213/ANE.0000000000000689. PMID 25822921
- [Derived] Welsby IJ, Schroeder DR, Ghadimi K, Nuttall GA, Smith MM. Thrombin generation after prothrombin complex concentrate or plasma transfusion during cardiac surgery. J Thromb Thrombolysis. 2025 Feb;58(2):309-318. doi: 10.1007/s11239-024-03061-3. Epub 2024 Dec 4. PMID 39633218
- [Derived] Hayes K, Fernando MC, Jordan V. Prothrombin complex concentrate in cardiac surgery for the treatment of coagulopathic bleeding. Cochrane Database Syst Rev. 2022 Nov 21;11(11):CD013551. doi: 10.1002/14651858.CD013551.pub2. PMID 36408876
- [Derived] Smith MM, Schroeder DR, Nelson JA, Mauermann WJ, Welsby IJ, Pochettino A, Montonye BL, Assawakawintip C, Nuttall GA. Prothrombin Complex Concentrate vs Plasma for Post-Cardiopulmonary Bypass Coagulopathy and Bleeding: A Randomized Clinical Trial. JAMA Surg. 2022 Sep 1;157(9):757-764. doi: 10.1001/jamasurg.2022.2235. PMID 35767271
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Fresh Frozen Plasma: After cardiopulmonary bypass, patients received protamine at dose 0.01 mg/unit of heparin given with target activated clotting time (ACT) within 10% of baseline value. After protamine administration the ACT, complete blood count (CBC), prothrombin time (PT)/ international normalized ratio (INR), activated partial thromboplastin time (APTT), and fibrinogen, were collected via preexisting arterial access. If ACT >10% baseline additional protamine was given at the anesthesiologists discretion. Evaluation and determination of excessive microvascular bleeding in the surgical field occurred 10 minutes after return of ACT to within 10% of baseline. Patients with clinical evidence of excessive microvascular bleeding in the surgical field as determined by the surgical team, along with a PT >16.6 sec/ INR >1.6 sec received fresh frozen plasma as this is standard therapy per our institutional algorithm at a dose of 10-15 mL/kg rounded up to the nearest unit.
  Fresh frozen plasma (FFP): FFP
- Prothrombin Complex Concentrate: After cardiopulmonary bypass, patients received protamine at dose 0.01 mg/unit of heparin given with target activated clotting time (ACT) within 10% of baseline value. After protamine administration the ACT, complete blood count (CBC), prothrombin time (PT)/ international normalized ratio (INR), activated partial thromboplastin time (APTT), and fibrinogen, were collected via preexisting arterial access. If ACT >10% baseline additional protamine was given at the anesthesiologists discretion. Evaluation and determination of excessive microvascular bleeding in the surgical field occurred 10 minutes after return of ACT to within 10% of baseline. Patients with clinical evidence of excessive microvascular bleeding in the surgical field as determined by the surgical team, along with a PT >16.6 sec/ INR >1.6 sec received Prothrombin complex concentrate (Human) 15 units/kg.
  Prothrombin complex concentrate (PCC) (Human): PCC (Kcentra)
Period: Overall Study
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate
Started | 53 | 53
Completed | 49 | 51
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Prothrombin Complex Concentrate: After cardiopulmonary bypass, patients received protamine at dose 0.01 mg/unit of heparin given with target activated clotting time (ACT) within 10% of baseline value. After protamine administration the ACT, complete blood count (CBC), prothrombin time (PT)/ international normalized ratio (INR), activated partial thromboplastin time (APTT), and fibrinogen, were collected via preexisting arterial access. If ACT >10% baseline additional protamine was given at the anesthesiologists discretion. Evaluation and determination of excessive microvascular bleeding in the surgical field occurred 10 minutes after return of ACT to within 10% of baseline. Patients with clinical evidence of excessive microvascular bleeding in the surgical field as determined by the surgical team, along with a PT >16.6 sec/ INR >1.6 sec received Prothrombin complex concentrate (Human) 15 units/kg.
  Prothrombin complex concentrate (Human): PCC (Kcentra)
- Total: Total of all reporting groups
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (14.6) | 68.1 (12.8) | 66.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 25 | 39
  Male | 35 | 26 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 50 | 98
  Hispanic or Latino | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Chest Tube Output
Description: The amount of chest tube drainage output from after surgery through midnight of the next day. As measured in mL.
Time Frame: 24 hours
Population: 1 subject's data was not collected nor analyzed for the FFP arm
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate
Number analyzed (Participants) | 48 | 51
mL | 1022 [799 to 1575] | 937 [708 to 1443]
Statistical Analysis 1: Comparison: Fresh Frozen Plasma vs Prothrombin Complex Concentrate; Test type: Superiority; p = 0.84, Regression, Linear; Ratio of the Geometric Means = 0.98, 95% CI 2-sided [0.81 to 1.19]

2. Primary Outcome: Red Blood Cell (RBC) Blood Product Transfusion
Description: The number of subject's who received 0,1,2,3 or more units of RBC's transfused from completion of study drug administration though midnight of the next day.
Time Frame: 24 hours
Population: 1 subject data was not collected nor analyzed for the FFP arm
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate
Number analyzed (Participants) | 48 | 51
Participants
  0 units | 26 | 36
  1 unit | 11 | 8
  2 units | 6 | 5
  3 or more units | 5 | 2
Statistical Analysis 1: Comparison: Fresh Frozen Plasma vs Prothrombin Complex Concentrate; Test type: Superiority; p = 0.09, Regression, Logistic; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.22 to 1.11]

3. Primary Outcome: Platelets Blood Product Transfusion
Description: The number of subject's who received 0,1,2,3 or more units of Platelets transfused from completion of study drug administration though midnight of the next day.
Time Frame: 24 hours
Population: 1 subject's data was not collected nor analyzed for the FFP arm
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate
Number analyzed (Participants) | 48 | 51
Participants
  0 units | 30 | 36
  1 unit | 13 | 9
  2 units | 3 | 3
  3 or more units | 2 | 3
Statistical Analysis 1: Comparison: Fresh Frozen Plasma vs Prothrombin Complex Concentrate; Test type: Superiority; p = 0.51, Regression, Logistic; Odds Ratio, log = 0.76, 95% CI 2-sided [0.33 to 1.73]

4. Primary Outcome: Cryoprecipitate (Cryo) Blood Product Transfusion
Description: The number of subject's who received 0,1,2,3 or more units of Cryo's transfused from completion of study drug administration though midnight of the next day.
Time Frame: 24 hours
Population: 1 subject's data was not collected nor analyzed for the FFP arm
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate
Number analyzed (Participants) | 48 | 51
Participants
  0 units | 40 | 40
  1 unit | 2 | 2
  2 units | 5 | 8
  3 or more units | 1 | 1
Statistical Analysis 1: Comparison: Fresh Frozen Plasma vs Prothrombin Complex Concentrate; Test type: Superiority; p = 0.53, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.51 to 3.79]

5. Primary Outcome: Fresh Frozen Plasma (FFP) Blood Product Transfusion
Description: The number of subject's who received 0,1,2,3 or more units of FFP's transfused from completion of study drug administration though midnight of the next day.
Time Frame: 24 hours
Population: 1 subject's data was not collected nor analyzed for the FFP arm
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate
Number analyzed (Participants) | 48 | 51
Participants
  0 units | 43 | 48
  1 unit | 0 | 1
  2 units | 4 | 2
  3 or more units | 1 | 0
Statistical Analysis 1: Comparison: Fresh Frozen Plasma vs Prothrombin Complex Concentrate; Test type: Superiority; p = 0.39, Regression, Logistic; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.12 to 2.30]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for each subject from baseline to end of study, approximately 30 days
Arm/Group | Fresh Frozen Plasma | Prothrombin Complex Concentrate
All-Cause Mortality (participants affected / at risk) | 2/49 | 1/51
Serious Adverse Events (participants affected / at risk) | 44/49 | 45/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fresh Frozen Plasma (N=49) | Prothrombin Complex Concentrate (N=51)
Anaphylactic or allergic reaction (Immune system disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 1
DVT (Vascular disorders) | 0 | 1
Mesenteric ischemia (Vascular disorders) | 3 | 1
Stroke/TIA (Nervous system disorders) | 1 | 2
STEMI (Cardiac disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 18 | 21
Renal Failure requiring dialysis (Renal and urinary disorders) | 4 | 5
ARDS (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Prolonged mechanical ventilation (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Re-operation (General disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT02557672/Prot_SAP_000.pdf